CLINICAL TRIAL: NCT00196313
Title: A Multicenter Study to Compare the Efficacy of an Extended-cycle Oral Contraceptive, Seasonique Which Utilizes Ethinyl Estradiol During the Usual Hormone-free Interval to Placebo for the Treatment of Cyclic Pelvic Pain in Adolescents
Brief Title: A Study to Evaluate the Efficacy of Seasonique for the Treatment of Cyclic Pelvic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR-PSE-306
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2012-05-25 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-08

CONDITIONS: Dysmenorrhea
Keywords: cyclic pelvic pain; dysmenorrhea; oral contraceptives
MeSH Terms: conditions — Dysmenorrhea | interventions — Seasonique

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 levonorgestrel/EE 0.15/0.03 and EE 0.01 mg tablet (Experimental)
  Interventions: Drug: levonorgestrel/EE 0.15/0.03 and EE 0.01 mg tablets
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: levonorgestrel/EE 0.15/0.03 and EE 0.01 mg tablets — 1 tablet daily by mouth
  Other Names: Seasonique
  Arms: 1 levonorgestrel/EE 0.15/0.03 and EE 0.01 mg tablet
Drug: Placebo tablet — 1 tablet daily by mouth
  Arms: 2

SUMMARY:
This study is being conducted to evaluate the effects of treatment with Seasonique an extended-regimen oral contraceptive that utilizes low dose ethinyl estradiol during the typical hormone-free interval. Patients will receive 13 weeks of treatment with the option to extend blinded therapy for an additional 13 weeks. The overall study duration will be 6-9 months. Patients will be required to record menstrual pain in a daily diary.

ELIGIBILITY:
Inclusion Criteria:

* Sexually naïve and agree to abstain from sex during the study
* Moderate to severe menstrual-related pelvic pain
* Regular spontaneous menstrual cycles

Exclusion Criteria:

* Any contraindication to the use of oral contraceptives
* Treatment with an oral contraceptive within the previous 3 months
* Previous treatment failure with an extended oral contraceptive regimen

Max Age: 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2005-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Duramed Investigational Site, Denver, Colorado
  - Duramed Investigational Site, Decatur, Georgia
  - Duramed Investigational Site, Louisville, Kentucky
  - Duramed Investigational Site, St Louis, Missouri
  - Duramed Investigational Site, Cincinnati, Ohio
  - Duramed Investigational Site, Cleveland, Ohio
  - Duramed Investigational Site, Columbus, Ohio
  - Duramed Investigational Site, Medford, Oregon
  - Duramed Investigational Site, Philadelphia, Pennsylvania
  - Duramed Investigational Site, Pittsburgh, Pennsylvania
  - Duramed Investigational Site, Willow Grove, Pennsylvania
  - Duramed Investigational Site, Providence, Rhode Island
  - Duramed Investigational Site, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 123 subjects were screened, of which 95 subjects were randomized. Of those randomized, 95 subjects took at lease 1 dose of study medication.
Groups:
- Seasonique: Seasonique
  , 1 tablet daily
- Placebo: Placebo, 1 tablet daily
Period: Overall Study
Arm/Group | Seasonique | Placebo
Started | 47 | 48
Completed | 36 | 40
Not Completed | 11 | 8
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Adverse Event | 3 | 1
Not completed — Subject Pregnant | 1 | 1
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Seasonique | Placebo | Total
Number analyzed (Participants) | 47 | 48 | 95
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.5 (1.23) | 15.4 (1.36) | 15.5 (1.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 48 | 95
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  African-American | 18 | 17 | 35
  Caucasian | 29 | 27 | 56
  Hispanic | 0 | 3 | 3
  Other | 0 | 1 | 1
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.8 (6.88) | 26.4 (7.16) | 25.6 (7.04)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Average Severity for Abdominal/Pelvic Pain
Description: Defined as the sum of pain scores divided by the total number of days in which the subject experienced abdominal/pelvic pain, from baseline to Week 13 The severity of the pain was assessed using a 4-points scale (0 = "None", 1 = "Mild", 2 = "Moderate", 3 = "Severe")
Time Frame: Baseline to end of 13-week treatment period
Population: Complete Cohort: consisted of all randomized subjects who completed the full term of study participation (13 weeks) and who had no recorded protocol violations that would have excluded the from analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Seasonique | Placebo
Number analyzed (Participants) | 36 | 40
units on a scale | -0.45 (0.060) | -0.19 (0.058)

2. Secondary Outcome: Change From Baseline in Maximum Severity of Abdominal/Pelvic Pain
Description: Maximum pain severity score was calculated by identifying each subject's maximum recorded pain severity from baseline to end of Week 13.
  The severity of the pain was assessed using a 4-points scale (0 = "None", 1 = "Mild", 2 = "Moderate", 3 = "Severe")
Time Frame: Baseline to end of Week 13
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Seasonique | Placebo
Number analyzed (Participants) | 36 | 40
units on a scale | -0.62 (0.120) | -0.17 (0.117)

3. Secondary Outcome: Incidence of Menstrual Bleeding and /or Spotting
Time Frame: Baseline to end of Week 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days of bleeding/spotting over 13 weeks
Groups:
- Seasonique: Seasonique, 1 tablet daily
Arm/Group | Seasonique | Placebo
Number analyzed (Participants) | 36 | 40
Days of bleeding/spotting over 13 weeks | 28.389 (14.705) | 18.000 (6.026)

4. Secondary Outcome: Number of Days Missed From School/Work or Other Activities
Time Frame: 13-week treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Seasonique | Placebo
Number analyzed (Participants) | 36 | 40
Days | 0.83 (1.844) | 2.75 (3.418)

5. Secondary Outcome: Analgesic Use
Description: number of days analgesic (pain) medication was used over the 13 week treatment period
Time Frame: 13-week treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days Analgesic was used over 13 weeks
Arm/Group | Seasonique | Placebo
Number analyzed (Participants) | 36 | 40
Days Analgesic was used over 13 weeks | 2.92 (3.281) | 4.03 (5.356)

ADVERSE EVENTS:
Arm/Group | Seasonique | Placebo
Serious Adverse Events (participants affected / at risk) | 2/47 | 0/48
Other Adverse Events (participants affected / at risk) | 47/47 | 17/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seasonique (N=47) | Placebo (N=48)
Excruciating pain rlated to menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Exacerbation of Stress (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seasonique (N=47) | Placebo (N=48)
Sinusitis (Infections and infestations) | 6 (6) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 5 (5)
Gastroenteritis Viral (Infections and infestations) | 4 (4) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (9) | 3 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 4 (4) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 9 (9) | 3 (3)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can (i) review results communications prior to public release and can embargo communications regarding trial results for a period of at least 60 days but no more than 180 days from the time submitted to the sponsor for review; and (ii) require in instances of a multi-center study, that a single PI not disclose study data until after the multi-center results are published, provided such results are published within eighteen (18) months of the conclusion of the study.